Distribution and Randomization of Gun Safety Devices to Measure Uptake and Preferences

NCT06682403 Unique Protocol ID: 855259

Document Date: 01/16/2024

Below is a voluntary survey that takes less than 3-minutes to complete.

After completing the survey, you will receive an Amazon gift card as compensation and be eligible to receive a free gun safety device shipped to your address.

Before you begin, please take a moment to review the consent form. If you have any questions or concerns, feel free to reach out to us at jane.maguire@pennmedicine.upenn.edu or Penn Medicine IRB at 215-898-2614.

- 1. The information shared in this survey will be used exclusively for research purposes and will be kept confidential.
- 2. The purpose of this survey is to better understand gun safety device preferences and storage use.
- 3. Participants' phone numbers will be used to deliver a digital Amazon gift card as a token of appreciation for survey completion and for re-contact with invitation to participate in the followup survey.
- 4. Your personal information will be stored securely. Your address will only be used as shipping information for the gun safety device.
- 5. You may stop the survey at any point without providing a reason.
- 6. Participation is totally voluntary, and you will not face any consequences for not participating.
- 7. The data from this survey will not be shared with anyone outside of the study team and will remain anonymous. The data will be used to inform future gun safety programs at Penn Medicine.
- 8. By selecting agree, you confirm that you've read and understand the items above and agree to participate in this survey and that you may be contacted for an opportunity to complete a follow-up survey.
- 9. By agreeing to participate in this survey, you acknowledge and agree that only one individual should complete the survey. We value the integrity of the survey responses provided. Any attempt to manipulate or falsify responses will result in disqualification of any associated payment.